CLINICAL TRIAL: NCT05171127
Title: Differentiation Between Healthy Cerebral Tissue and Tumor Tissue Using a Tissue Sensing Instrument
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Oscar Persson, MD, PhD, Karolinska University Hospital
Other Study IDs: 2019-00100
Record Dates: First submitted 2021-12-11; First posted 2021-12-28 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Glioblastoma; Surgical Margin
MeSH Terms: conditions — Glioblastoma; Margins of Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glioblastoma: No intervention. Observation of diffuse reflectance spectroscopy patterna are made on ex-vivo tissue samples in patients undergoing surgery for glial tumors.
  Interventions: Procedure: Diffuse Reflectance Spectroscopy

INTERVENTIONS:
Procedure: Diffuse Reflectance Spectroscopy — Measurements of DRS patterns in extirpated tumor and cerebral tissue

SUMMARY:
Differentiation between glioma tumor tissue and normal cerebral tissue using Diffuse Reflectance Spectroscopy (DRS) on surgical tissue samples ex-vivo

DETAILED DESCRIPTION:
Background: Diffuse reflectance spectroscopy is an optically based technique which measures the amount of diffusely reflected light after it has undergone multiple scattering and absorption events within the tissue. Each DRS spectrum therefore has a specific 'optical fingerprint' reflecting the composition and morphology of the tissue within the probing volume. The technology is easily built into very small instruments that can be fused with regularly used surgical equipment. DRS has previously been widely investigated for the purpose of margin assessment in other regions of the body.

Aim & Hypothesis: The primary goal is to show the feasibility of applying optical tissue sensing using diffuse reflectance spectroscopy (DRS) to differentiate healthy cerebral tissue from tumorous tissue in ex vivo human tissue samples. This will be a basis for further development of surgical equipment able to identify the margin between healthy brain tissue and tumor tissue intraoperatively.

Method: Using DRS we aim to determine spectroscopy thresholds that enables differentiation of cerebral tissue from different forms of tumor tissue. We aim to determine these thresholds by collecting DRS data on ex vivo brain and tumor samples. The tumor samples will be part of the normal extraction of tissue during tumor surgeries and the non tumorous tissue can be extracted in temporal/frontal lobe resections as well as epilepsy surgery, where non tumorous brain tissue is to be removed. The DRS measurements are performed in direct connection to the extraction of tissue during surgery, and the tissue is thereafter sent to the pathologist according to standard clinical procedures. No extra tissue will need to be resected for the purpose of this study. Based on the experiments we will propose a theoretical model for differentiating normal cerebral tissue from tumor tissue in humans for use during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical resection of glial tumor or epileptic focus

Exclusion Criteria:

* Unable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing surgical resection of glial tumors or non-neoplastic cerebral lesions at Karolinska University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
DRS pattern | simultaneously with surgery
  Diffuse Reflectance Spectroscopy pattern in tissue type

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Persson, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No